CLINICAL TRIAL: NCT04397172
Title: Characterization of ARDS, Critical Illness Myopathy and Their Long-term Consequences in Patients With Covid-19 Disease: Effects of Inflammation, Mitochondrial Dysfunction and Plasma Concentrations of Various Sedative Drugs
Brief Title: Intensive Care Associated Complications and Outcome of Acute Respiratory Distress Syndrome Due to COVID-19
Status: Terminated | Type: Observational
Why Stopped: Number of Covid-19 cases who need intensive care have greatly reduced, it is very difficult to find eligible patients for the study
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00730
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: COVID; Corona Virus Infection; Sars-CoV2
Keywords: Corona; SARS-CoV2; ARDS; PICS
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Study Arm — First inpatient examination (within 24 hours after admission to ICU):
  * Clinical examination
  * Laboratory tests, Biobanking, Mitochondrial function testing
  * Neurophysiological examination (MVRC recording)
  Follow-up inpatient examinations (day 2, 5 and 10 after admission):
  * Clinical examination
  * Laboratory tests, Biobanking, Mitochondrial functions testing
  * Neurophysiological examination (MVRC recording)
  * Day 10 only: Extended neurophysiological examination according to diagnostic criteria
  * Day 10 only: Grading of muscle strength (Medical Research Council (MRC) system)
  Follow-up outpatient examination (after discharge from intensive care):
  * Clinical examination
  * Grading of muscle strength (MRC)
  * Modified Rankin Scale (mRS)
  * Barthel Scale
  * Questionnaires (Short Form (36) Health Survey, Essener Questionnaire for Coping with a Disease and Beck's Depression Inventory II)

SUMMARY:
COVID-19 patients with a severely symptomatic progression with development of an Acute respiratory distress syndrome (ARDS) due to SARS-CoV-2 need prolonged intensive care treatment involving pharmacological immobilization, sedation and mechanical ventilation, leaving them at a very high risk for developing Critical illness myopathy (CIM). CIM is associated with increased mortality and significant consequences for recovery and the ability to return to normal daily life. Up to date, there are no studies investigating the mid- or long-term course of the novel COVID-19 disease. The present study therefore aims to evaluate the clinical outcome of patients with ARDS due to SARS-CoV-2 with special attention to the development of CIM and its underlying causes. To provide the possibility of early diagnosis of CIM, critically ill patients will be regularly screened for muscle membrane alterations using (Muscle velocity recovery cycles) MRVC measurements.

The primary endpoint is the incidence of CIM in patients with ARDS due to SARS-CoV-2, diagnosed according to the current diagnostic criteria.

DETAILED DESCRIPTION:
COVID-19 patients with a severely symptomatic progression with development of an ARDS due to SARS-CoV-2 need prolonged intensive care treatment involving pharmacological immobilization, sedation and mechanical ventilation, leaving them at a very high risk for developing CIM. CIM is associated with increased mortality and significant consequences for recovery and the ability to return to normal daily life. Up to date, there are no studies investigating the mid- or long-term course of the novel COVID-19 disease. The present study therefore aims to evaluate the clinical outcome of patients with ARDS due to SARS-CoV-2 with special attention to the development of CIM and its underlying causes. To provide the possibility of early diagnosis of CIM, critically ill patients will be regularly screened for muscle membrane alterations using MRVC measurements.

Objective:

The primary objective of this project is to prospectively evaluate the incidence and severity of CIM in patients with ARDS due to SARS-CoV-2.

The secondary objectives of this project include:

1. To assess the quality of life of patients with and without CIM after ARDS due to SARS-CoV-2.
2. To monitor changes in muscle excitability parameters in critically ill patients with ARDS due to SARS-CoV-2 in relation to a later confirmed diagnosis of CIM according to the current standards.
3. To explore underlying pathophysiological processes for CIM (mitochondrial dysfunction, medication e.g. Neuromuscular blocking agents (NMBA), sedative drugs, and metabolic (amino acids, inflammatory parameters)).

Method:

After enrolment in the study, patients will be examined for the first time within 24 hours after admission to the ICU, and follow-up visits will be performed at day 2, 5 and 10 or upon termination of therapy with NMBA, respectively. The endpoint will be at the clinical follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by a surrogate assessment by an independent physician
* Adult ICU Patients with ARDS due to SARS-CoV-2 requiring mechanical ventilation

Exclusion Criteria:

* Age <18 years and > 80 years
* Pregnancy and breast feeding
* The presence of pre-existing:

  * Known (at time of inclusion) Polyneuropathy,
  * Known (at time of inclusion) Guillain-Barré syndrome,
  * Known (at time of inclusion) Acute or chronic spinal cord lesion,
  * Known (at time of inclusion) Myasthenia gravis, or
  * Known (at time of inclusion) Myopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study aims to prospectively evaluate the incidence and severity of CIM in patients with ARDS due to SARS-CoV-2.
  The investigators therefore conduct a study including patients with ARDS admitted to the intensive care unit (ICU) due to the novel COVID-19 disease (SARS-CoV-2). The investigators plan to analyze 50 full data sets of ICU patients (regarding primary endpoint), out of which about 30-50% will be expected to develop CIM. There is no alternative group of patients with whom this study could be conducted.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Short Form (36) Health Survey (SF-36) | 3 months
  Short Form (36) Health Survey (SF-36)

SECONDARY OUTCOMES:
Mortality | 90 days
  Mortality
Modified Rankin Scale (mRS) | 90 days
  Modified Rankin Scale (mRS); (0=no Symptoms at all, 6=dead)
Duration of mechanical ventilation in days | 3 months
  Duration of mechanical ventilation in days
Barthel Index | 3 months
  Barthel Index (80-100= patient should be able to live independently, <20=total dependence)
Beck's Depression Inventory II (BDI-II) | 3 months
  Beck's Depression Inventory II (BDI-II)
Essener Questionnaire for Coping with a Disease (EFK) | 3 months
  Essener Questionnaire for Coping with a Disease (EFK); (0=no burden of disease, 180-strong burden of disease)
Number of patients with Critical Illness Myopathy | day 10
  Number of patients with Critical Illness Myopathy

CONTACTS AND LOCATIONS:
Overall Officials: Werner Z'Graggen, MD, Principal Investigator — Universitätsklinik für Neurochirurgie und Neurologie
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belgnaoui SM, Paz S, Hiscott J. Orchestrating the interferon antiviral response through the mitochondrial antiviral signaling (MAVS) adapter. Curr Opin Immunol. 2011 Oct;23(5):564-72. doi: 10.1016/j.coi.2011.08.001. Epub 2011 Aug 22. PMID 21865020
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Dinglas VD, Aronson Friedman L, Colantuoni E, Mendez-Tellez PA, Shanholtz CB, Ciesla ND, Pronovost PJ, Needham DM. Muscle Weakness and 5-Year Survival in Acute Respiratory Distress Syndrome Survivors. Crit Care Med. 2017 Mar;45(3):446-453. doi: 10.1097/CCM.0000000000002208. PMID 28067712
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] de Letter MA, Schmitz PI, Visser LH, Verheul FA, Schellens RL, Op de Coul DA, van der Meche FG. Risk factors for the development of polyneuropathy and myopathy in critically ill patients. Crit Care Med. 2001 Dec;29(12):2281-6. doi: 10.1097/00003246-200112000-00008. PMID 11801825
- [Background] Griffiths J, Hatch RA, Bishop J, Morgan K, Jenkinson C, Cuthbertson BH, Brett SJ. An exploration of social and economic outcome and associated health-related quality of life after critical illness in general intensive care unit survivors: a 12-month follow-up study. Crit Care. 2013 May 28;17(3):R100. doi: 10.1186/cc12745. PMID 23714692
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] James MA. Use of the Medical Research Council muscle strength grading system in the upper extremity. J Hand Surg Am. 2007 Feb;32(2):154-6. doi: 10.1016/j.jhsa.2006.11.008. No abstract available. PMID 17275587
- [Background] Lacomis D. Electrophysiology of neuromuscular disorders in critical illness. Muscle Nerve. 2013 Mar;47(3):452-63. doi: 10.1002/mus.23615. Epub 2013 Feb 6. PMID 23386582
- [Background] Latronico N, Bolton CF. Critical illness polyneuropathy and myopathy: a major cause of muscle weakness and paralysis. Lancet Neurol. 2011 Oct;10(10):931-41. doi: 10.1016/S1474-4422(11)70178-8. PMID 21939902
- [Background] Liu Y, Yan LM, Wan L, Xiang TX, Le A, Liu JM, Peiris M, Poon LLM, Zhang W. Viral dynamics in mild and severe cases of COVID-19. Lancet Infect Dis. 2020 Jun;20(6):656-657. doi: 10.1016/S1473-3099(20)30232-2. Epub 2020 Mar 19. No abstract available. PMID 32199493
- [Background] Shi CS, Qi HY, Boularan C, Huang NN, Abu-Asab M, Shelhamer JH, Kehrl JH. SARS-coronavirus open reading frame-9b suppresses innate immunity by targeting mitochondria and the MAVS/TRAF3/TRAF6 signalosome. J Immunol. 2014 Sep 15;193(6):3080-9. doi: 10.4049/jimmunol.1303196. Epub 2014 Aug 18. PMID 25135833
- [Background] Weber-Carstens S, Deja M, Koch S, Spranger J, Bubser F, Wernecke KD, Spies CD, Spuler S, Keh D. Risk factors in critical illness myopathy during the early course of critical illness: a prospective observational study. Crit Care. 2010;14(3):R119. doi: 10.1186/cc9074. Epub 2010 Jun 18. PMID 20565863
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Z'Graggen WJ, Brander L, Tuchscherer D, Scheidegger O, Takala J, Bostock H. Muscle membrane dysfunction in critical illness myopathy assessed by velocity recovery cycles. Clin Neurophysiol. 2011 Apr;122(4):834-41. doi: 10.1016/j.clinph.2010.09.024. Epub 2010 Nov 1. PMID 21044861